







## **ARC Provider Information and Consent Form-Interview**

<u>Title of Study</u>: ARC – Access to Resources in the Community

Principal Investigator (PI) Simone Dahrouge, PhD 613-562-6262 ext. 2913 **Funding Agencies**:

Canadian Institutes of Health Research SPOR initiative

Participation in this study is voluntary. Please read this Informed Consent Form carefully before you decide if you will take part. You may also ask the study team as many questions as you like.

#### Why am I being invited to do an interview?

Your practice and you are participants in a research study about improving access to community resources for patients; the Access to Resources in the Community (ARC) study. Some primary care providers participating in that study are being invited to participate in an interview at the end of the study to understand their experience with the intervention.

#### What should I expect in participating in this interview?

The interview would be at a time and place that is convenient for you. It may be done by phone or face to face, depending on your preference.

You will be asked to answer some questions regarding your experience with the study. For example, the study team would like to understand whether you felt that the Patient Navigator's role was appropriate, and whether you felt that your patients have benefitted from that support.

The interview will take about 30 minutes. With your permission, the discussion will be audio recorded to ensure we have properly captured your answers. If you do not want to be audio recorded, you can still participate in the interview.

#### What are the risks involved in taking part in this interview?

There are minimal risks. You might find the interview is long or that the questions feel personal. You might not like all of the questions that you are asked. You do not have to answer any questions that make you uncomfortable.

#### Can I expect to benefit from participating in this interview?

You may not directly benefit from your participation in the interview; however, your participation may help the researchers to better understand the value of the Patient Navigator, and can potentially help future patients in getting more suitable support.

### How is my personal information being protected?

Your personal information will be protected just as it will be in the main study. The interview files will be identified by a study participant ID only and not by any information that may identify you such as your name. The link between your participant ID and name will be kept securely and separately from the study data.

If you agree to be audiotaped the audio recordings will be sent to a professional to produce a written document of the interview. Any information that could identify you, such as your name, will be removed from the transcription. Only the study team and the professional producing the written document of the







interview will have access to the audio recording and written form of the interview, and data will only be identified by a study ID. Study data will be kept by the study team for ten years – this is the same for all studies. After ten years, your information will be safely deleted or destroyed.

### Do I have to take part in this interview?

The decision to take part in the interview is entirely up to you. The decision to participate or not will not influence your participation in the ARC study.

You can refuse to answer any question during the interview.

If you choose to participate and change your mind, you may withdraw at any time, and if you wish, all the information that you have provided will be removed and will not be used in the study.

Your decision to participate in this study or not will <u>not</u> impact your employment status within your practice.

#### Who do I contact if I have any further questions?

If you have any questions about this study, please email us (arc@bruyere.org).

The Ottawa Health Science Network Research Ethics Board (OHSN-REB), the Bruyère Research Ethics Board, the Hôpital Montfort Research Ethics Board, and the University of Ottawa Research Ethics Board have reviewed this protocol. These Boards consider the ethical aspects of all research studies involving human participants at participating hospitals, institutes and universities.

If you have any questions about your rights as a study participant, you may contact:

- Chairperson, OHSN-REB at 613-798-5555, ext. 16719
- Research Ethics Coordinator, Bruyère Research Ethics Board at <u>reb@bruyere.org</u> or 613-562-6262 ext. 4003.
- Chairperson, Hôpital Montfort Research Ethics Board at 613-746-4111 ext. 6402
- Protocol Officer for Ethics in Research, University of Ottawa, <u>at ethics@uottawa.ca</u> or 613-562-5387
- Research Ethics Officer, Laurentian University at 705-675-1151 ext 3213, 2436 or toll free at 1-800-461-4030 or email ethics@laurentian.ca.
- Ethics and Compliance Officer, University of Ontario Institute of Technology, researchethics@uoit.ca or 905-721-8668 X 3693

Should you no longer wish to remain a part of the ARC study, please call Andrea Perna (613) 562-6262 ext.2920 or email <u>arc@bruyere.org</u>. In Sudbury, please call Patrick Timony (705) 675-1151 ext. 4298 or email Pe Timony@laurentian.ca

You can also contact the study principal investigator, Simone Dahrouge at (613) 562-6262 ext. 2913 or sdahrouge@bruyere.org. In Sudbury, please contact Alain Gauthier at (705) 675-1151 ext: 4301 or email agauthier@laurentian.ca



# Access to Resources in the Community

# **Consent to Participate in an Interview**

| <ul> <li>I understand that I am being asked to take part in an interview at the end<br/>about my experience with the study.</li> </ul> | of the ARC study to talk |
|---|---|
| • has explained the process to me. | |
| I read each page of this form, or had this form read to me. | |
| All of my questions were answered so that I understand the study. | |
| • I can decide at any time that I do not want to take part in this interview. | |
| I have decided to take part in this interview. | |
| • I will get a copy of this signed form. | |
| I agree to have my interview audio recorded. | |
| Participant's Printed Name (Provider) Provider Signature | Date |
| Investigator or Delegate Statement I have carefully explained the study to the participant. To the best of my kunderstands the nature, demands, risks and benefits involved in taking part in to the lateral demands and benefits involved in taking part in the lateral demands. Investigator/Delegate's Printed Name Investigator/Delegate's Signature | chis study. |
| 5 | |